CLINICAL TRIAL: NCT06651957
Title: The Relationship Between Anal High-Risk HPV (Hr-HPV) Infection, Anal High-Grade Squamous Intraepithelial Lesions (HSIL), and the Anal Microbiome Among Three Distinct Populations of Hispanic People Living With HIV (PLWH) in California, Mexico and Puerto Rico
Brief Title: Anal High-risk HPV, HSIL, and Microbiome Among Hispanic Peoples Living With HIV (PLWH)
Acronym: ULACNet-104
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 24361; NCI-2024-01760 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); U54CA242646 (NIH)
Record Dates: First submitted 2024-10-18; First posted 2024-10-22 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Human Immunodeficiency Virus; Human Papillomavirus-Related Anal Squamous Cell Carcinoma; High-Grade Squamous Intraepithelial Lesions
Keywords: Microbiome
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Squamous Intraepithelial Lesions | interventions — Specimen Handling; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Anal swabs will be obtained for analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Participants undergo collection of 3 anal swab samples, complete questionnaires, and have their medical records reviewed on study. Participants with visible lesions undergo non-investigational high resolution anoscope with a non-investigational anal biopsy per usual care on study.
  Interventions: Other: Biospecimen Collection; Other: Questionnaires

INTERVENTIONS:
Other: Biospecimen Collection — Specimen swabs will be obtained.
  Other Names: Specimen Collection
Other: Questionnaires — Given to participants
  Other Names: Study-related questionnaires

SUMMARY:
The study evaluates if there is relationship between the kinds of bacteria living in the anus (also known as the anal microbiome) and the risk of human papillomavirus (HPV) infection or HPV-related pre-cancer (high-grade squamous intraepithelial lesions or HSIL) in Hispanic people living with HIV (PLWH) in Puerto Rico, Mexico and California

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Study the relationship between anal high-risk HPV (hr-HPV) infection and the anal microbiome among three distinct populations of Hispanic people living with HIV (PLWH) in Mexico, Puerto Rico, and California.

OUTLINE:

This is an observational study.

Participants undergo collection of 3 anal swab samples, complete questionnaires, and have their medical records reviewed on study. Participants with visible lesions undergo high resolution anoscope with anal biopsy per usual care on study.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of HIV-1 infection by means of any one of the following:

  * Documentation of HIV diagnosis in the medical record by a licensed health care provider.
  * Documentation of receipt of antiretroviral therapy (ART) by a licensed health care provider (Documentation may be a record of an ART prescription in the participant's medical record, a written prescription in the name of the participant for ART, or pill bottles for ART with a label showing the participant's name. Receipt of at least two agents is required; each component agent of a multi-class combination ART regimen will be counted toward the 2-agent requirement, excepting receipt of a pre-exposure prophylaxis (PrEP) regimen alone (e.g., Truvada), which is exclusionary);
  * HIV-1 RNA detection by a licensed HIV-1 RNA assay demonstrating >1000 RNA copies/mL;
  * Any locally licensed HIV screening antibody and/or HIV antibody/antigen combination assay confirmed by a second licensed HIV assay such as a HIV-1 Western blot confirmation or HIV rapid multispot antibody differentiation assay.
  * NOTE: A "licensed" assay refers to a U.S. FDA-approved assay or an assay approved by the relevant local health authority.
* Age 21 years or older. Cervical HSIL/cancer screening does not usually begin until 20 years of age or older. Also, anal HSIL/cancer screening among high-risk individuals such as people living with HIV is recommended for those 25 years of age or older. Children under the age of 18 are at low risk of developing cervical or anal HSIL/cancer and will not benefit from the kind of screening planned for this study.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 (Karnofsky score ≥ 70%).
* Ability to understand and the willingness to sign a written informed consent document.
* Previous consent to participate in ULACNet-101 in Mexico and Puerto Rico sites or a patient at Anal Neoplasia Clinic, Research and Education (ANCRE) Center in San Francisco.

Exclusion Criteria:

* History of inflammatory bowel disease or colorectal cancer
* Participants with active evidence of proctitis.
* Participants on immunosuppressive drugs. Exclusion criteria from ULACNet-101
* Participants who have undergone hysterectomy.
* History of anal cancer, penile, vulvar, vaginal, or cervical cancer.
* Potential participants who received prior treatment of anal, cervical, penile, vaginal, or vulvar lesions within 18 months of study enrollment.
* Inability, in the opinion of the study investigator, of the participant to comply with study requirements.
* Participants who are pregnant (a urine pregnancy test will be provided to participants of age 60 years or less) or within 2 months postpartum.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hispanic participants previously consented to ULACNet-101 study diagnosed with HIV and received antiretroviral therapy
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Evaluate association between with hr-HPV and pro-inflammatory-mediating taxa | Up to 1 year
  Among Hispanic PLWH without anal high-grade squamous intraepithelial lesions (HSIL), the investigators hypothesize the microbiome will be different between those with and without hr-HPV infection and the proportion with pro-inflammatory-mediating taxa will be highest among the Puerto Rican population compared with the Mexican and California populations given the higher incidence in anal cancer in Puerto Rico.
Association between with hr-HPV and butyrate-producing signatures | Up to 1 year
  Among Hispanic PLWH with anal hr-HPV at the three locations, the investigators hypothesize the detection of HSIL will be associated with a pro-inflammatory microbiome and a decrease in butyrate-producing signatures, with the proportion of pro-inflammatory changes highest among the Puerto Rican population compared with the Mexican and California populations.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Palefsky, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- University of California, San Francisco, San Francisco, California, United States
- Instituto Nacional de Salud Publica, Cuernavaca, Morelos, Mexico
- University of Puerto Rico, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with research collaborators
Supporting Information: Study Protocol

DOCUMENTS (1):
  • Informed Consent Form (2025-02-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT06651957/ICF_000.pdf